CLINICAL TRIAL: NCT06784765
Title: Preventive Use of Pressurized Intraperitoneal Aerosol Chemotherapy in Locally Advanced Gastric Cancer: A Non-Randomized Controlled Study
Brief Title: Preventive Use of PIPAC in Locally Advanced Gastric Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Oncology and Transplantology Center, Kazakhstan (Other)
Collaborators: Ministry of Science and Higher Education of the Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Altay Kerimkulov, MD, Principal investigator, National Research Oncology and Transplantology Center, Kazakhstan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAZNEOPAC; BR24992950 (Other Grant/Funding Number: Committee of Science of the Ministry of Science and Higher Education of the Republic of Kazakhstan)
Record Dates: First submitted 2024-12-31; First posted 2025-01-20 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; peritoneal carcinomatosis; gastrectomy; PIPAC; FLOT
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Doxorubicin; Cisplatin; Gastrectomy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PIPAC+FLOT (Experimental): ◦ Preventive pressurized intraperitoneal aerosol chemotherapy (PIPAC) with cisplatin (10 mg/m2) and doxorubicin (2.1 mg/m2) + perioperative chemotherapy (FLOT regimen) + gastrectomy with D2 D2 lymphadenectomy.
  Interventions: Procedure: Intervention Group
- FLOT (Active Comparator): Retrospective cohort receiving standard perioperative chemotherapy (FLOT regimen) + gastrectomy with D2 D2 lymphadenectomy.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Intervention Group — Preventive pressurized intraperitoneal aerosol chemotherapy (PIPAC) with cisplatin (10 mg/m2) and doxorubicin (2.1 mg/m2) + perioperative chemotherapy (FLOT regimen) +gastrectomy with D2 lymphadenectomy
  Other Names: doxorubicin (2.1 mg/m2); cisplatin (10 mg/m2); perioperative chemotherapy (FLOT regimen); gastrectomy; D2 lymphadenectomy; Preventive pressurized intraperitoneal aerosol chemotherapy (PIPAC)
  Arms: PIPAC+FLOT
Procedure: Control Group — Retrospective cohort receiving standard perioperative chemotherapy (FLOT regimen) + gastrectomy with D2 lymphadenectomy
  Other Names: standard perioperative chemotherapy (FLOT regimen); gastrectomy; D2 lymphadenectomy
  Arms: FLOT

SUMMARY:
Gastric cancer is the fifth most common cancer worldwide and the third leading cause of cancer-related mortality. In patients with locally advanced gastric cancer, multimodal treatment strategies, including perioperative chemotherapy, have significantly improved survival rates. Despite these advances, peritoneal carcinomatosis (PC) remains a serious problem, occurring in 60% of cases after radical surgery. PC is associated with poor prognosis and limited treatment options.

Intra-abdominal chemotherapy, particularly hyperthermic intraperitoneal chemoperfusion (HIPEC), has demonstrated advantages in the treatment of PC. However, a new technique, pressurized intraperitoneal aerosolized chemotherapy (PIPAC), is emerging as a promising alternative. PIPAC delivers chemotherapeutic agents directly to the peritoneal surface as an aerosol, allowing deeper penetration of drugs into tumor implants while minimizing toxicity and invasiveness.

This study hypothesizes that the addition of PIPAC as a preoperative treatment for patients with locally advanced gastric cancer may reduce the incidence of peritoneal carcinomatosis compared to standard therapy. The primary objective of this study is to determine whether preoperative PIPAC reduces the incidence of peritoneal carcinomatosis in these patients.

DETAILED DESCRIPTION:
Gastric cancer is the fifth most common cancer globally and the third leading cause of cancer-related death. In patients with locally advanced gastric cancer, multimodal treatment strategies, including perioperative chemotherapy, have significantly improved survival outcomes. However, PC remains a major challenge, often occurring in 60% of cases after radical surgery, and is associated with a poor prognosis and limited treatment options.

Intra-abdominal chemotherapy, particularly HIPEC, has shown benefits in the treatment of PC. However, a newer method, PIPAC, is emerging as a promising alternative. PIPAC delivers chemotherapeutic agents directly to the peritoneal surface via aerosol, ensuring deeper penetration of the drugs into tumor implants and offering lower toxicity and less invasiveness compared to traditional methods.

This study hypothesizes that adding PIPAC as a preoperative treatment in patients with locally advanced gastric cancer may reduce the occurrence of peritoneal carcinomatosis compared to standard therapy alone. PIPAC will be applied before neoadjuvant chemotherapy to patients at high risk for peritoneal recurrence, with the goal of improving survival rates and reducing recurrence after surgery.

The main objectives of this study are to determine whether preoperative PIPAC reduces the incidence of peritoneal carcinomatosis in patients with locally advanced gastric cancer. Secondary objectives include assessing overall survival (OS), progression-free survival (PFS), disease-free survival (DFS), the occurrence of serious adverse events (SAEs), quality of life (QoL) as measured by the EORTC QLQ-C30, postoperative mortality (Clavien-Dindo classification), and pathological response (TRG) in comparison to patients receiving standard treatment.

ELIGIBILITY:
Adults aged 18-70 years with histologically confirmed locally advanced gastric adenocarcinoma (T3-4N0-3M0), ECOG performance status 0-2, and negative peritoneal cytology.

Inclusion Criteria:

1. Signed informed consent
2. Aged 18-70 years
3. ECOG performance status 0-2
4. Histologically confirmed adenocarcinoma of the stomach (T3-4N0-3M0)
5. Negative peritoneal cytology from diagnostic laparoscopy
6. No prior chemotherapy or radiotherapy

Exclusion Criteria:

1. Presence of distant metastases
2. Positive peritoneal cytology
3. Previous cancer treatment (chemotherapy, radiotherapy, or surgery)
4. Severe comorbid conditions contraindicating surgery or chemotherapy
5. Pregnancy or lactation
6. Known hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of peritoneal carcinomatosis | 12, 24 months after surgery
  Incidence of Peritoneal Carcinomatosis refers to the frequency or rate at which new cases of peritoneal carcinomatosis are diagnosed within a specific population over a defined period.

SECONDARY OUTCOMES:
Overall survival | 1. 3, 5 years after surgery
  Overall Survival (OS) refers to the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients are still alive.
Disease-free survival | 3, 6, 9, 12, 18, 24 months after surgery
  Disease-Free Survival (DFS) is the period of time after treatment during which a patient shows no signs of the disease.
Quality of life by EORTC QLQ-C30 | before surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  Quality of life (assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), which is calculated in points)
Frequency of adverse events | through study completion, 30 days after surgery, 90 days after surgery
  Frequency of Adverse Events (graded by CTCAE v5.0) refers to the rate or proportion of patients experiencing side effects or complications associated with a treatment, categorized according to severity using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Oncology Centre, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sgarbura O, Eveno C, Alyami M, Bakrin N, Guiral DC, Ceelen W, Delgadillo X, Dellinger T, Di Giorgio A, Kefleyesus A, Khomiakov V, Mortensen MB, Murphy J, Pocard M, Reymond M, Robella M, Rovers KP, So J, Somashekhar SP, Tempfer C, Van der Speeten K, Villeneuve L, Yong WP, Hubner M. Consensus statement for treatment protocols in pressurized intraperitoneal aerosol chemotherapy (PIPAC). Pleura Peritoneum. 2022 Mar 1;7(1):1-7. doi: 10.1515/pp-2022-0102. eCollection 2022 Mar 1. PMID 35602919
- [Background] Coccolini F, Nardi M, Montori G, Ceresoli M, Celotti A, Cascinu S, Fugazzola P, Tomasoni M, Glehen O, Catena F, Yonemura Y, Ansaloni L. Neoadjuvant chemotherapy in advanced gastric and esophago-gastric cancer. Meta-analysis of randomized trials. Int J Surg. 2018 Mar;51:120-127. doi: 10.1016/j.ijsu.2018.01.008. Epub 2018 Feb 20. PMID 29413875
- [Background] Al-Batran SE, Lorenzen S. Management of Locally Advanced Gastroesophageal Cancer: Still a Multidisciplinary Global Challenge? Hematol Oncol Clin North Am. 2017 Jun;31(3):441-452. doi: 10.1016/j.hoc.2017.01.004. Epub 2017 Mar 29. PMID 28501086
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Background] Cotte E, Passot G, Gilly FN, Glehen O. Selection of patients and staging of peritoneal surface malignancies. World J Gastrointest Oncol. 2010 Jan 15;2(1):31-5. doi: 10.4251/wjgo.v2.i1.31. PMID 21160814
- [Derived] Kerimkulov A, Uskenbayev T, Sarina T, Mamlin M, Shalekenov S, Yessenbayeva G, Kainazarov T, Burkitbayev Z, Ussipbekov B, Kovalchuk D, Rakhmankulov A, Rakhmankulova A, Gaipov A. Efficacy of Preventive Pressurized Intraperitoneal Aerosol Chemotherapy in Patients With Locally Advanced Gastric Cancer: Protocol for a Prospective Controlled Trial. JMIR Res Protoc. 2025 Nov 11;14:e78053. doi: 10.2196/78053. PMID 41218205